CLINICAL TRIAL: NCT02916381
Title: The Analgesic Efficacy of the Pectoral Block After Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, PD Dr, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 2016-01413
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEC block (Experimental): Ultrasound-guided PEC block after induction of general anaesthesia.
  Interventions: Procedure: PEC block + General anaesthesia
- Control (Sham Comparator): No ultrasound-guided PEC block; only general anaesthesia will be provided.
  Interventions: Procedure: General anaesthesia

INTERVENTIONS:
Procedure: PEC block + General anaesthesia — Patients will receive an ultrasound-guided PEC block after the induction of general anaesthesia.
  Arms: PEC block
Procedure: General anaesthesia
  Arms: Control

SUMMARY:
Unilateral mastectomy is associated with moderate to severe postoperative pain. A new regional anaesthetic technique has been recently described, call the PEC block. This technique consists of injecting local anaesthetic between different muscles of the chest in order to relieve postoperative pain. The investigators aim to verify that this technique has a clinical relevant postoperative analgesic effect. For that purpose, the investigators will randomise 50 patients scheduled to undergo unilateral mastectomy into two groups: one group will receive a PEC block after the induction of the general anaesthesia under ultrasound guidance, while the other group will not have this regional procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Age ≥ 18
* Patients undergoing unilateral mastectomy

Exclusion Criteria:

* Contraindications to regional block
* Pregnancy
* Inability to give informed consent
* History of alcohol or drug dependence/abuse
* History of long term opioid intake or chronic pain disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Intravenous morphine consumption during the first 24 postoperative hours (mg) | Postoperative day 1

SECONDARY OUTCOMES:
Intravenous morphine consumption on postoperative day 2 (mg) | Postoperative day 2
Intravenous morphine consumption in phase 1 recovery (mg) | 2 postoperative hours
Pain scores at rest in phase 1 recovery (visual analogue scale, 0 - 10) | 2 postoperative hours
  (visual analogue scale, 0 - 10)
Pain scores at rest on postoperative day 1 (visual analogue scale, 0 - 10) | Postoperative day 1
  Visual analogue scale, 0 - 10)
Pain scores at rest on postoperative day 2 (visual analogue scale, 0 - 10) | Postoperative day 2
  Visual analogue scale, 0 - 10)
Postoperative nausea and vomiting (yes/no) | Postoperative day 1
Postoperative nausea and vomiting (yes/no) | Postoperative day 2
Pruritus (yes/no) | Postoperative day 1
Pruritus (yes/no) | Postoperative day 2

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, Principal Investigator — CHUV
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland